CLINICAL TRIAL: NCT07324018
Title: Efficacy of a Spirulina Derivative in Preventing Radiation-Induced Esophagitis in Esophageal Cancer Patients Undergoing IMRT: A Randomized Controlled Trial
Brief Title: Spirulina Derivative for Radiation Esophagitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025(2393)
Record Dates: First submitted 2025-12-03; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Radiation-induced Esophagitis
Keywords: esophageal cancer; radiation-induced esophagitis; spirulina; exosome
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogel of placebo (Placebo Comparator)
  Interventions: Drug: Hydrogel of placebo; Radiation: Radiotherapy
- Hydrogel of spirulina derivatives (Experimental)
  Interventions: Drug: Hydrogel of spirulina-derived exosomes.; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Hydrogel of spirulina-derived exosomes. — An oral hydrogel formulated with purified spirulina-derived exosomes.
  Arms: Hydrogel of spirulina derivatives
Drug: Hydrogel of placebo — The placebo oral hydrogel will be formulated with inactive ingredients matched in appearance and flavor profile to the active spirulina-derived product.
  Arms: Hydrogel of placebo
Radiation: Radiotherapy — Patient eligibility was defined as a diagnosis of esophageal cancer with a treatment plan involving radiotherapy (radiotherapy alone or concurrent chemoradiotherapy) using intensity-modulated radiotherapy (IMRT).

SUMMARY:
To evaluate the efficacy and safety of a Spirulina-derived product in preventing and treating radiation-induced esophagitis in esophageal cancer patients undergoing intensity-modulated radiotherapy (IMRT).

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of a spirulina-derived product in reducing the incidence, duration, and severity of radiation-induced esophagitis in esophageal cancer patients. The study primarily aims to address two questions: (1) whether the spirulina-derived product can effectively prevent and mitigate radiation-induced esophageal injury, and (2) whether its use is associated with adverse events in patients undergoing intensity-modulated radiotherapy (IMRT).

Participants will be instructed to orally administer the spirulina-derived product or placebo solution four times daily, starting from the first day of radiotherapy and continuing throughout the RT course. After each administration, patients must refrain from eating, drinking, or performing oral intake for at least 1 hour to maximize mucosal contact time of the intervention.

The study will compare the spirulina-derived product group with the placebo group to determine the potential benefits of this spirulina-based intervention in preventing and managing radiotherapy-related esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histopathologically confirmed malignant esophageal tumor and no distant metastasis;
2. Age ≥ 18 years;
3. ECOG (Eastern Cooperative Oncology Group) performance status score ≤ 2;
4. Scheduled to undergo definitive radiotherapy, neoadjuvant radiotherapy, or adjuvant radiotherapy for esophageal cancer;
5. Adequate hepatic, renal, and bone marrow function;
6. Signed informed consent form.

Exclusion Criteria:

1. History of prior thoracic radiotherapy.
2. Known allergy to spirulina or its derivatives, any component of the thermosensitive gel, or having a history of severe allergic predisposition.
3. Presence of esophageal or oral diseases assessed by the investigator before radiotherapy initiation that may affect the analysis of this study's results (e.g., reflux esophagitis, Barrett's esophagus, severe oral infection, recurrent aphthous ulcers, oral lichen planus, etc.).
4. Use of systemic antibacterial or antifungal medications within one week prior to the start of radiotherapy.
5. Planned concurrent use of medications that may exacerbate radiation-induced mucosal injury after radiotherapy initiation (e.g., anti-EGFR monoclonal antibodies, immune checkpoint inhibitors, etc.).
6. Presence of severe underlying diseases of the cardiovascular, pulmonary, hepatic, renal, hematopoietic, or nervous systems (specific criteria for organ dysfunction are detailed in item 7 below), or conditions such as acute infection, uncontrolled autoimmune diseases, poorly controlled diabetes mellitus, etc., which, in the investigator's judgment, may increase study risks or interfere with result analysis.
7. Presence of significant organ dysfunction meeting any of the following criteria:

   * Hemoglobin < 80 g/L;
   * Neutrophil count < 1.0 × 10⁹/L;
   * Platelet count < 80 × 10⁹/L;
   * Serum total bilirubin ≥ 2 times the upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 times ULN;
   * Serum creatinine > 1.5 times ULN.
8. Pregnant or lactating women.
9. History of severe mental illness, alcohol abuse, or drug abuse.
10. Participation in other clinical trials within the past 3 months.
11. Any other condition deemed by the investigator as potentially rendering the subject unsuitable for participation in this study (e.g., extremely poor oral hygiene, poor compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥2 radiation-induced esophagitis (RTOG criteria). | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks to 14.5 weeks.
  Radiation esophagitis is assessed by trained radiotherapists according to the Radiation Therapy Oncology Group (RTOG) acute radiation morbidity scoring criteria. The RTOG criteria categorize acute esophageal toxicity into grades 0-4, with a higher grade indicating more severe symptoms. Grade 0 represents no change over baseline; grade 1 represents mild dysphagia or odynophagia requiring topical anesthetic or non-narcotic analgesics/soft diet; grade 2 represents moderate dysphagia or odynophagia requiring narcotic analgesics/pureed or liquid diet; grade 3 represents severe dysphagia or odynophagia with dehydration or weight loss (>15% from pre-treatment baseline) requiring nasogastric feeding tube, intravenous fluids, or hyperalimentation; and grade 4 represents complete obstruction, ulceration, perforation, or fistula formation.

SECONDARY OUTCOMES:
Duration of Grade ≥2 Radiation Esophagitis | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  Toxicity Monitoring: Radiation oncologists or research nurses, uniformly trained, will assess and record the specific grade of esophagitis in patients at predefined time points, strictly adhering to the RTOG Acute Radiation Morbidity Scoring Criteria.
  Start Point Determination: The date when esophagitis is first recorded as grade ≥2 during the observation period is defined as the start date of the toxicity event.
  End Point Determination: The date when esophagitis is first recorded as having decreased and subsequently maintained at grade 1 or 0 in follow-up assessments is defined as the end date (i.e., recovery date) of the toxicity event.
  Duration Calculation: The duration of a single event is calculated as: End Date - Start Date. If the patient's esophagitis grade has not decreased to grade 0 by the end of the observation period (8 weeks after radiotherapy completion), the duration data for that patient will be treated as censored data.
Time to Onset of Grade ≥2 Esophagitis | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  Toxicity Monitoring: Radiation oncologists or research nurses, uniformly trained, will assess and record the specific grade of esophagitis in patients at predefined time points, strictly adhering to the RTOG Acute Radiation Morbidity Scoring Criteria.
  Onset Point Determination: The date when esophagitis is first recorded as grade ≥2 during the observation period is defined as the onset date of this toxicity event.
  Assessment Time Window: From the start of radiotherapy until 8 weeks after radiotherapy completion. To accurately capture the timing of toxicity onset, assessments are planned twice weekly during radiotherapy and once weekly during the follow-up period after radiotherapy completion.
  Handling of Special Cases: If a patient has not experienced grade ≥2 esophagitis by the end of the observation period (8 weeks post-radiotherapy), the time data for this endpoint will be treated as censored data.
Adverse events | From the start of radiotherapy to 8 weeks after completion of radiotherapy.The evaluation period is approximately 14 weeks to 14.5 weeks.
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version

OTHER OUTCOMES:
The longitudinal dynamics of salivary microbiota | From the start of radiotherapy (baseline) to treatment completion. The total evaluation period is approximately 6 to 6.5 weeks.
  Measurement Description: This indicator assesses the dynamic changes in the composition (relative abundance of microbial taxa) and alpha diversity (e.g., Shannon index, Chao1 index) of the salivary microbiota in cancer patients undergoing radiotherapy throughout the treatment process.
  Measurement Methods:
  Sample Collection: Non-stimulated whole saliva samples are collected from patients at specified time points using the spit method.
  Laboratory Analysis: Total microbial DNA is extracted from the saliva samples. The V3-V4 hypervariable regions of the bacterial 16S rRNA gene are amplified via PCR, followed by sequencing using the Illumina high-throughput sequencing platform.
  Bioinformatics Analysis: Raw sequencing data undergo quality control, denoising, and generation of amplicon sequence variants. These are then aligned and annotated against reference databases to analyze the community structure and diversity of the microbiota.
Overall Health Status and Core Dimensions of Quality of Life | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) This instrument is a 30-item patient-reported outcome (PRO) measure designed to evaluate core aspects of health-related quality of life in cancer patients, including 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, pain, nausea and vomiting), one global health status/quality of life scale, and 6 single-item symptom measures. Scores are linearly transformed to a range of 0-100. For the functional scales and the global health status scale, higher scores indicate better functional levels or quality of life; for the symptom scales/items, higher scores indicate greater symptom burden.
Esophageal Cancer-Specific Symptoms | From the start of radiotherapy (baseline) to 2 months after treatment completion. The total evaluation period is approximately 14 to 14.5 weeks.
  Description of Measurement Method:
  The EORTC QLQ-OES18 is a patient-reported outcome (PRO) instrument specifically designed to assess disease-related symptoms and treatment-related side effects in patients with esophageal cancer. It comprises 18 items, organized into four multi-item subscales (dysphagia, eating, reflux, and pain) and six single-item measures (dry mouth, taste problems, coughing, speech problems, difficulty swallowing saliva, and hair loss). All subscale and single-item scores are linearly transformed to a 0-100 scale using a standardized scoring algorithm.
  Interpretation of Scores:
  For all subscales and single items, higher scores represent more severe symptoms or greater symptom burden.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No